CLINICAL TRIAL: NCT02725879
Title: Association of Serum Fibroblast Growth Factor 21 (FGF-21) Levels With Resting Metabolic Rate (RMR), in Children and Adolescents With Hashimoto's Thyroiditis.
Brief Title: FGF-21 Levels and RMR in Children and Adolescents With Hashimoto's Thyroiditis (THYROMETABOL)
Acronym: THYROMETABOL
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Assimina Galli-Tsinopoulou, Professor, Aristotle University Of Thessaloniki
Other Study IDs: PEDIATRIC ENDOCRINOLOGY
Record Dates: First submitted 2016-01-09; First posted 2016-04-01 (Estimated); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hashimoto Disease
Keywords: fibroblast growth factor 21; resting metabolic rate; chronic autoimmune thyroiditis; L-thyroxin; children; adolescents
MeSH Terms: conditions — Hashimoto Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- AIT Subclinical Hypothyroid Group: 30 children and adolescents with subclinical hypothyroidism due to Hashimoto's thyroiditis.
  No special intervention is to be administered, only routine LT4 treatment. Reassessment at 6 months.
- Control Group: 30 healthy individuals with no chronic autoimmune thyroiditis and normal thyroid function (age- and sex-matched with the AIT Subclinical Hypothyroid Group).
  No special intervention is to be administered. No reassessment at 6 months.
- AIT Euthyroid Group: 30 children and adolescents with chronic autoimmune thyroiditis and euthyroidism (age- and sex-matched with the AIT Subclinical Hypothyroid Group).
  No special intervention is to be administered. No reassessment at 6 months.

SUMMARY:
It is well documented that thyroid hormones (THs) are involved in energy and lipid metabolism, thermogenesis, and body weight control, acting on several tissues. Thus, any change in thyroid status may affect body weight and metabolic rate. On the other hand, fibroblast growth factor 21 (FGF-21) is a complex hormone involved in energy, lipid, and glucose metabolism, sharing common biochemical pathways and sites of action with THs. FGF-21 is synthesized and acts primarily on the liver, but weaker expression has also been described in muscle, pancreas, and adipose tissue. In addition, FGF-21 acts through endocrine and paracrine mechanisms, regulating metabolic pathways such as fatty acid oxidation, glucose uptake, and thermogenesis. Recent animal and human studies have highlighted a close bidirectional relationship between FGF-21 and THs, partially elucidated. Thyroid hormones regulate the expression of the FGF-21 gene in the liver and can also increase FGF-21 levels in vivo. However, it has also been suggested that some of their key actions are largely independent. Data on FGF-21 levels and their metabolic role in pediatric patients with chronic autoimmune thyroiditis (AIT) are scarce. This study aims to measure FGF-21 serum levels in children and adolescents with Hashimoto's thyroiditis and investigate any possible associations between FGF-21 serum levels and resting metabolic rate (RMR) and levothyroxine (LT4) treatment, or other clinical and biochemical parameters.

DETAILED DESCRIPTION:
Children and adolescents, aged 5-18 years, will undergo routine screening for chronic autoimmune thyroiditis (AIT) at the Pediatric Endocrinology Outpatient Clinic of "Papageorgiou" General Hospital and "AHEPA" University Hospital of Thessaloniki, Greece. The diagnosis of AIT will be based on the presence of anti-thyroid autoantibodies (Anti-TPOAb and/or Anti-TgAb) and one or more of the following: clinical symptoms of thyroid dysfunction, goiter, or diffuse/irregular hypoechogenicity of the thyroid gland during an ultrasound examination.

All participants should have a normal body mass index (BMI) for their age and sex, be drug-naive for at least 3 months, follow no special diet, and have no chronic and/or acute disease or menstrual disorder. Only those subjects that will start routine LT4 treatment will be reassessed at six months (not the rest participants), with no specific intervention to take place during those six months.

For all participants, a detailed medical history will be recorded. The following parameters will be measured and calculated: age and pubertal stage according to Tanner, height, body weight, Body Mass Index (BMI), waist circumference, hip circumference, mid-upper arm circumference (MUAC), and skinfolds measurement in order to estimate the percentage of body fat (%BF). The resting metabolic rate (RMR) will be measured with a portable device applying indirect calorimetry. Blood samples will be collected after overnight fasting.

The following parameters will be tested in serum: thyroid-stimulating hormone (TSH), free triiodothyronine (FT3), free thyroxine (FT4), anti-thyroid peroxidase antibody (Anti-TPOAb) titers, thyroglobulin antibody (Anti-TgAb) titers, total cholesterol (TC), triglyceride (TG), high-density lipoprotein (HDL), low-density lipoprotein (LDL), aspartate aminotransferase (AST), alanine aminotransferase (ALT), γglutamyltransferase (γ-GT), alkaline phosphatase (ALP), applying an automatic chemical analyzer or immunoassay system and analogs reagents that already exist at the hospital. Serum FGF-21 levels will be determined in pg/mL using the Solid Phase Sandwich Enzyme-linked Immunosorbent Assay (ELISA) method according to the manufacturer's protocol.

Additionally, all participants, with the help of their parents and/or caregivers, will complete the Mediterranean Diet Index (KIDMED) at their first visit.

ELIGIBILITY:
Inclusion Criteria:

For patients

* Subjects 5 to 18 years old.
* First diagnosis of chronic autoimmune thyroiditis (high levels of serum antithyroid autoantibodies anti-TPO, anti-TgAb).

For Controls:

* Healthy individuals 5 to 18 years old.
* BMI for age between 15th and 85th percentile (z-score between -1 and +1).

Exclusion Criteria:

For patients

* Pre-existing medical treatment for thyroid disease
* Taking other medications (eg growth hormone, corticosteroids) in the last 3 months.
* Taking food supplements (eg omega-3 fatty acids, amino acids) in the last 3 months.
* Concomitant endocrine, metabolic, degenerative, and/or chronic diseases other than obesity (eg diabetes, hyper/ hypercortisolemia, cardiovascular diseases, kidney diseases, myasthenia, neurological diseases, psychiatric disorders eg anorexia nervosa, cancer, anemia, celiac disease, chromosomal abnormalities eg syndrome Turner, Down, etc).
* Participation in any daily organized physical activity (sport), more than 1 hour per day.
* Presence of menstrual disorders in adolescent girls.
* Having any kind of nutrition/dietary intervention (eg weight loss diet, hypocaloric, ketogenic, low-protein diet), in the last 6 months.

For Controls:

* Presence of any form of thyroid disease.
* Presence of any endocrine, metabolic, degenerative, and/or chronic disease (eg diabetes, hyper/ hypercortisolemia, obesity, metabolic syndrome, cardiovascular diseases, kidney diseases, myasthenia, neurological diseases, psychiatric disorders eg anorexia nervosa, cancer, anemia, celiac disease, chromosomal abnormalities eg syndrome Turner, Down, etc).
* Taking any medication (eg growth hormone, corticosteroids) in the last 3 months.
* Taking food supplements (eg omega-3 fatty acids, amino acids) in the last 3 months.
* Participation in any daily organized physical activity (sport), more than 1 hour per day. Presence of menstrual disorders in adolescent girls.
* Having any kind of nutrition/dietary intervention (eg weight loss diet, hypocaloric, ketogenic, low-protein diet), in the last 6 months.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and Adolescents of Greek origin who attend the Pediatric Endocrinology Outpatient Units of 4th and 2nd Departments of Pediatrics, Medical School, Aristotle University of Thessaloniki for testing thyroid autoimmunity, as well as healthy controls.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Assimina Galli-Tsinopoulou, MD,PhD, Principal Investigator — 2nd Department of Paediatrics, AΗEPA Hospital
Locations (1):
- 2nd Department of Paediatrics, School of Medicine Faculty of Health Sciences, Aristotle University of Thessaloniki, AHEPA Hospital Thessaloniki, Greece, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams AC, Astapova I, Fisher FM, Badman MK, Kurgansky KE, Flier JS, Hollenberg AN, Maratos-Flier E. Thyroid hormone regulates hepatic expression of fibroblast growth factor 21 in a PPARalpha-dependent manner. J Biol Chem. 2010 May 7;285(19):14078-82. doi: 10.1074/jbc.C110.107375. Epub 2010 Mar 17. PMID 20236931
- [Background] Astrup A, Buemann B, Toubro S, Ranneries C, Raben A. Low resting metabolic rate in subjects predisposed to obesity: a role for thyroid status. Am J Clin Nutr. 1996 Jun;63(6):879-83. doi: 10.1093/ajcn/63.6.879. PMID 8644681
- [Background] Barbesino G, Chiovato L. The genetics of Hashimoto's disease. Endocrinol Metab Clin North Am. 2000 Jun;29(2):357-74. doi: 10.1016/s0889-8529(05)70136-5. PMID 10874534
- [Background] Coskun T, Bina HA, Schneider MA, Dunbar JD, Hu CC, Chen Y, Moller DE, Kharitonenkov A. Fibroblast growth factor 21 corrects obesity in mice. Endocrinology. 2008 Dec;149(12):6018-27. doi: 10.1210/en.2008-0816. Epub 2008 Aug 7. PMID 18687777
- [Background] Dayan CM, Daniels GH. Chronic autoimmune thyroiditis. N Engl J Med. 1996 Jul 11;335(2):99-107. doi: 10.1056/NEJM199607113350206. No abstract available. PMID 8649497
- [Background] Dostalova I, Kavalkova P, Haluzikova D, Lacinova Z, Mraz M, Papezova H, Haluzik M. Plasma concentrations of fibroblast growth factors 19 and 21 in patients with anorexia nervosa. J Clin Endocrinol Metab. 2008 Sep;93(9):3627-32. doi: 10.1210/jc.2008-0746. Epub 2008 Jun 17. PMID 18559909
- [Background] Griffiths M, Payne PR, Stunkard AJ, Rivers JP, Cox M. Metabolic rate and physical development in children at risk of obesity. Lancet. 1990 Jul 14;336(8707):76-8. doi: 10.1016/0140-6736(90)91592-x. PMID 1975323
- [Background] Hanks LJ, Casazza K, Ashraf AP, Wallace S, Gutierrez OM. Fibroblast growth factor-21, body composition, and insulin resistance in pre-pubertal and early pubertal males and females. Clin Endocrinol (Oxf). 2015 Apr;82(4):550-6. doi: 10.1111/cen.12552. Epub 2014 Aug 8. PMID 25039824
- [Background] Iglesias P, Selgas R, Romero S, Diez JJ. Biological role, clinical significance, and therapeutic possibilities of the recently discovered metabolic hormone fibroblastic growth factor 21. Eur J Endocrinol. 2012 Sep;167(3):301-9. doi: 10.1530/EJE-12-0357. Epub 2012 Jun 27. PMID 22740503
- [Background] Kim KH, Lee MS. FGF21 as a Stress Hormone: The Roles of FGF21 in Stress Adaptation and the Treatment of Metabolic Diseases. Diabetes Metab J. 2014 Aug;38(4):245-51. doi: 10.4093/dmj.2014.38.4.245. PMID 25215270
- [Background] Lee P, Linderman JD, Smith S, Brychta RJ, Wang J, Idelson C, Perron RM, Werner CD, Phan GQ, Kammula US, Kebebew E, Pacak K, Chen KY, Celi FS. Irisin and FGF21 are cold-induced endocrine activators of brown fat function in humans. Cell Metab. 2014 Feb 4;19(2):302-9. doi: 10.1016/j.cmet.2013.12.017. PMID 24506871
- [Background] Lee Y, Park YJ, Ahn HY, Lim JA, Park KU, Choi SH, Park DJ, Oh BC, Jang HC, Yi KH. Plasma FGF21 levels are increased in patients with hypothyroidism independently of lipid profile. Endocr J. 2013;60(8):977-83. doi: 10.1507/endocrj.ej12-0427. Epub 2013 Jun 12. PMID 23759753
- [Background] Mai K, Schwarz F, Bobbert T, Andres J, Assmann A, Pfeiffer AF, Spranger J. Relation between fibroblast growth factor-21, adiposity, metabolism, and weight reduction. Metabolism. 2011 Feb;60(2):306-11. doi: 10.1016/j.metabol.2010.02.016. Epub 2010 Apr 1. PMID 20362303
- [Background] McAninch EA, Bianco AC. Thyroid hormone signaling in energy homeostasis and energy metabolism. Ann N Y Acad Sci. 2014 Apr;1311:77-87. doi: 10.1111/nyas.12374. Epub 2014 Feb 20. PMID 24697152
- [Background] Mraz M, Bartlova M, Lacinova Z, Michalsky D, Kasalicky M, Haluzikova D, Matoulek M, Dostalova I, Humenanska V, Haluzik M. Serum concentrations and tissue expression of a novel endocrine regulator fibroblast growth factor-21 in patients with type 2 diabetes and obesity. Clin Endocrinol (Oxf). 2009 Sep;71(3):369-75. doi: 10.1111/j.1365-2265.2008.03502.x. Epub 2008 Dec 11. PMID 19702724
- [Background] Muller TD, Tschop MH. Play down protein to play up metabolism? J Clin Invest. 2014 Sep;124(9):3691-3. doi: 10.1172/JCI77508. Epub 2014 Aug 18. PMID 25133420
- [Background] Nakamura MT, Yudell BE, Loor JJ. Regulation of energy metabolism by long-chain fatty acids. Prog Lipid Res. 2014 Jan;53:124-44. doi: 10.1016/j.plipres.2013.12.001. Epub 2013 Dec 18. PMID 24362249
- [Background] Pyrzak B, Demkow U, Kucharska AM. Brown Adipose Tissue and Browning Agents: Irisin and FGF21 in the Development of Obesity in Children and Adolescents. Adv Exp Med Biol. 2015;866:25-34. doi: 10.1007/5584_2015_149. PMID 26022904
- [Background] Santini F, Marzullo P, Rotondi M, Ceccarini G, Pagano L, Ippolito S, Chiovato L, Biondi B. Mechanisms in endocrinology: the crosstalk between thyroid gland and adipose tissue: signal integration in health and disease. Eur J Endocrinol. 2014 Oct;171(4):R137-52. doi: 10.1530/EJE-14-0067. PMID 25214234
- [Background] Skarpa V, Kousta E, Tertipi A, Anyfandakis K, Vakaki M, Dolianiti M, Fotinou A, Papathanasiou A. Epidemiological characteristics of children with autoimmune thyroid disease. Hormones (Athens). 2011 Jul-Sep;10(3):207-14. doi: 10.14310/horm.2002.1310. PMID 22001131
- [Background] Vaidya B, Kendall-Taylor P, Pearce SH. The genetics of autoimmune thyroid disease. J Clin Endocrinol Metab. 2002 Dec;87(12):5385-97. doi: 10.1210/jc.2002-020492. No abstract available. PMID 12466323
- [Background] Woelnerhanssen B, Peterli R, Steinert RE, Peters T, Borbely Y, Beglinger C. Effects of postbariatric surgery weight loss on adipokines and metabolic parameters: comparison of laparoscopic Roux-en-Y gastric bypass and laparoscopic sleeve gastrectomy--a prospective randomized trial. Surg Obes Relat Dis. 2011 Sep-Oct;7(5):561-8. doi: 10.1016/j.soard.2011.01.044. Epub 2011 Mar 22. PMID 21429816
- [Background] Xu J, Lloyd DJ, Hale C, Stanislaus S, Chen M, Sivits G, Vonderfecht S, Hecht R, Li YS, Lindberg RA, Chen JL, Jung DY, Zhang Z, Ko HJ, Kim JK, Veniant MM. Fibroblast growth factor 21 reverses hepatic steatosis, increases energy expenditure, and improves insulin sensitivity in diet-induced obese mice. Diabetes. 2009 Jan;58(1):250-9. doi: 10.2337/db08-0392. Epub 2008 Oct 7. PMID 18840786
- [Background] Zhang A, Sieglaff DH, York JP, Suh JH, Ayers SD, Winnier GE, Kharitonenkov A, Pin C, Zhang P, Webb P, Xia X. Thyroid hormone receptor regulates most genes independently of fibroblast growth factor 21 in liver. J Endocrinol. 2015 Mar;224(3):289-301. doi: 10.1530/JOE-14-0440. Epub 2014 Dec 11. PMID 25501997

RESULTS

PARTICIPANT FLOW:
Groups:
- AIT Subclinical Hypothyroid Group: Children and Adolescents diagnosed with chronic autoimmune thyroiditis (AIT) and subclinical hypothyroidism (SCH), who received standard levothyroxine (LT4) treatment.
- Control Group: Healthy individuals with no chronic autoimmune thyroiditis (AIT) and normal thyroid function (age- and sex-matched with AIT Treatment Group).
- AIT Euthyroid Group: Children and Adolescents diagnosed with chronic autoimmune thyroiditis (AIT) and euthyroidism (age- and sex-matched with AIT Subclinical Hypothyroid Group).
Period: Overall Study
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Started | 30 | 30 | 30
Completed | 30 | 30 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: AIT Subclinical Hypothyroid group: diagnosed with chronic autoimmune thyroiditis (AIT) and subclinical hypothyroidism (SCH), receiving standard levothyroxine (LT4) treatment.
  Control group: Healthy, no chronic autoimmune thyroiditis (AIT) and normal thyroid function (age- and sex-matched with AIT Subclinical Hypothyroid Group).
  AIT Euthyroid group: diagnosed with chronic autoimmune thyroiditis (AIT) and euthyroidism (age- and sex-matched with AIT Subclinical Hypothyroid Group).
Groups:
- AIT Subclinical Hypothyroid Group: Children and Adolescents diagnosed with chronic autoimmune thyroiditis (AIT) and subclinical hypothyroidism (SCH), receiving standard levothyroxine (LT4) treatment.
- Control Group: Healthy individuals with no chronic autoimmune thyroiditis (AIT) and normal thyroid function (age- and sex-matched with AIT Subclinical Hypothyroid Group).
- Total: Total of all reporting groups
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 30 | 30 | 90
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.99 (1.85) | 10.89 (2.29) | 11.01 (1.93) | 10.97 (2.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 18 | 54
  Male | 12 | 12 | 12 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 30 | 30 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 30 | 30 | 30 | 90
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Fibroblast Growth Factor 21 (FGF-21)
Description: serum fibroblast growth factor 21 (FGF-21) levels after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" at the 6 month time point. Data have not been collected for the "AIT Euthyroid Group" for the baseline and 6 month time points.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- AIT Subclinical Hypothyroid Group: Children and Adolescents diagnosed with chronic autoimmune thyroiditis (AIT) and subclinical hypothyroidism (SCH) , receiving standard levothyroxine (LT4) treatment.
- AIT Euthyroid Group: Children and Adolescents with chronic autoimmune thyroiditis and euthyroidism (age- and sex-matched with AIT Subclinical Hypothyroid Group).
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 0
pg/mL
  baseline | 182.71 [169.32 to 234.55] | 217.36 [193.60 to 235.21] |
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 198.43 [183.86 to 248.42] |  |

2. Primary Outcome: RMR/Weight/Day
Description: Resting Metabolic Rate (RMR) per kilogram of body weight per day
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: kJ/kg/day
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
kJ/kg/day
  baseline | 131.08 [108.62 to 165.10] | 150.46 [122.09 to 190.58] | 168.74 [133.26 to 193.51]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 142.51 [116.61 to 168.53] |  |

3. Secondary Outcome: SDS BMI
Description: Standard Deviation Score (SDS) for Body Mass Index (BMI). The standard deviation is a measure of the amount of variation or spread of a set of values around the mean or average. The mean or average value is given an SDS of "0". A negative SDS indicates that the value is below the average or mean and a positive value means it is above the average or mean. SDS correspond to growth chart percentiles as follow:
  -2.68 = 0.4th percentile, -2.01 = 2nd percentile, -1.34 = 9th percentile, -0.67 = 25th percentile, 0 (mean or average) = 50th percentile, +0.67 = 75th percentile, +1.34 = 91st percentile, +2.01 = 98th percentile, +2.68 = 99.6th percentile.
  These percentiles help us understand whether a measurement falls within the normal range for children of the same age and sex. A lower SDS value (closer or lower to -2.68) and a higher SDS value (closer or above +2.68) mean a worst outcome, while a SDS value closer to 0 (mean or average), mean a better outcome.
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
score on a scale
  baseline | 0.73 [0.12 to 1.64] | 0.88 [-0.01 to 1.22] | 0.36 [-1.07 to 1.16]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 0.88 [0.10 to 1.50] |  |

4. Secondary Outcome: WAIST C.
Description: Waist Circumference
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
cm
  baseline | 67.73 (9.32) | 69.33 (9.99) | 65.65 (8.59)
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 69.2 (8.61) |  |

5. Secondary Outcome: HIP C.
Description: Hip circumference
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
cm
  baseline | 81.38 (9.58) | 80.63 (10.58) | 77.41 (9.69)
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 81.50 (14.71) |  |

6. Secondary Outcome: MUAC
Description: mid-upper arm circumference
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
cm
  baseline | 22.00 [20.00 to 25.25] | 23.00 [20.00 to 25.25] | 21.00 [19.75 to 23.62]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 23.00 [22.00 to 26.00] |  |

7. Secondary Outcome: %BF
Description: Body fat percentage (%BF), is the total mass of fat divided by total body mass. The total body fat includes essential body fat and stored body fat.
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: percentage of body fat
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
percentage of body fat
  baseline | 24.95 [21.15 to 32.07] | 22.6 [18.53 to 31.8] | 21.65 [16.47 to 29.83]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 24.06 [19.27 to 31.16] |  |

8. Secondary Outcome: FMI
Description: Fat mass index (FMI) is calculated by dividing the fat weight in kilograms by the height in metres squared.
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
kg/m^2
  baseline | 4.49 [3.43 to 7.06] | 4.42 [3.17 to 5.98] | 4.12 [2.64 to 5.63]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 8.98 [4.87 to 13.4] |  |

9. Secondary Outcome: FFMI
Description: Fat free mass index (FFMI) is calculated by dividing the free fat weight in kilograms by the height in metres squared.
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
kg/m^2
  baseline | 14.27 [13.50 to 14.63] | 14.66 [13.43 to 15.31] | 13.47 [12.69 to 14.58]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 24.90 [18.52 to 31.31] |  |

10. Secondary Outcome: TSH
Description: thyroid-stimulating hormone (TSH) after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: μIU/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
μIU/L
  baseline | 4.82 [3.99 to 9.66] | 2.40 [1.95 to 3.06] | 2.63 [2.13 to 3.09]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 4.03 [2.43 to 6.20] |  |

11. Secondary Outcome: FT3
Description: free triiodothyronine after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
pmol/L
  baseline | 5.96 [5.44 to 6.44] | 6.28 [5.71 to 6.79] | 6.27 [5.91 to 6.71]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 5.90 [5.22 to 6.21] |  |

12. Secondary Outcome: FT4
Description: free thyroxine (FT4) after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
pmol/L
  baseline | 14.29 (2.45) | 15.19 (1.93) | 15.19 (2.57)
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 15.70 (2.45) |  |

13. Secondary Outcome: Glucose
Description: glucose serum level after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
mmol/L
  baseline | 4.86 [4.66 to 5.12] | 4.88 [4.65 to 5.11] | 4.74 [4.49 to 5.05]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 4.97 [4.72 to 5.19] |  |

14. Secondary Outcome: Insulin
Description: insulin serum level after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
pmol/L
  baseline | 64.58 [46.46 to 86.87] | 48.12 [37.36 to 81.32] | 54.65 [33.96 to 81.87]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 65.07 [47.85 to 87.43] |  |

15. Secondary Outcome: TC
Description: Total Cholesterol (TC) serum level after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
mmol/L
  baseline | 4.22 (0.84) | 3.88 (0.75) | 4.22 (0.69)
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 4.19 (0.86) |  |

16. Secondary Outcome: TG
Description: Triglyceride (TG) serum level after an overnight fasting
Time Frame: baseline and 6 month
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
mmol/L
  baseline | 0.74 [0.52 to 0.89] | 0.52 [0.45 to 0.65] | 0.66 [0.56 to 1.02]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 0.73 [0.56 to 0.93] |  |

17. Secondary Outcome: HDL
Description: high-density lipoprotein (HDL) serum level after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
mmol/L
  baseline | 1.43 [1.18 to 1.65] | 1.38 [1.23 to 1.63] | 1.54 [1.24 to 1.99]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 1.46 [1.26 to 1.61] |  |

18. Secondary Outcome: LDL
Description: low-density lipoprotein (LDL) serum level after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
mmol/L
  baseline | 2.30 [2.01 to 2.92] | 2.07 [1.65 to 2.56] | 2.33 [2.04 to 2.64]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 2.30 [1.93 to 2.82] |  |

19. Secondary Outcome: AST
Description: aspartate aminotransferase (AST) serum level after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
IU/L
  baseline | 23.00 [19.00 to 25.25] | 24.50 [18.75 to 28.25] | 27.50 [23.75 to 29.00]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 22.00 [18.00 to 25.00] |  |

20. Secondary Outcome: ALT
Description: alanine aminotransferase (ALT) serum level after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
IU/L
  baseline | 15.00 [13.00 to 19.50] | 14.50 [13.00 to 18.00] | 16.50 [13.75 to 19.00]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 15.50 [13.75 to 19.25] |  |

21. Secondary Outcome: γ-GT
Description: gamma gloutamyltransferase (γ-GT) serum level after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
IU/L
  baseline | 12.00 [10.75 to 15.00] | 12.00 [10.00 to 13.25] | 12.00 [11.00 to 13.25]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 11.00 [10.00 to 14.00] |  |

22. Secondary Outcome: ALP
Description: alkaline phosphatase (ALP) serum level after an overnight fasting
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
IU/L
  baseline | 200.00 [157.75 to 291.50] | 217 [149.5 to 275.50] | 217.00 [183.25 to 275.00]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 224.50 [162.50 to 270.25] |  |

23. Secondary Outcome: Homeostatic Model Assessment for Insulin Resistance (HOMA-IR)
Description: HOMA-IR stands for Homeostatic Model Assessment of Insulin Resistance, using fasting insulin and blood glucose levels after an overnight fastιng. The meaningful part of the acronym is "insulin resistance". It marks for both the presence and extent of any insulin resistance that you might currently express. It is a way to reveal the dynamic between the baseline (fasting) blood sugar and the responsive hormone insulin.
  Healthy Range: 1.0 (0.5-1.4) Less than 1.0 means you are insulin-sensitive which is optimal. Above 1.9 indicates early insulin resistance. Above 2.9 indicates significant insulin resistance.
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the 6 month time point.
Measure: Median (Inter-Quartile Range); unit: index
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
index
  baseline | 1.93 [1.39 to 2.72] | 1.50 [1.11 to 2.54] | 1.62 [1.02 to 2.52]
  6 months: number analyzed (Participants) | 30 | 0 | 0
  6 months | 1.90 [1.57 to 2.65] |  |

24. Secondary Outcome: Mediterranean Diet Index (KIDMED) Score
Description: Mediterranean diet index (KIDMED) score is a questionnaire used to evaluate adherence to the Mediterranean diet in children and adolescents. The KIDMED assesses how well an individual's dietary habits align with the Mediterranean diet.
  Scoring System: 16 questions, each associated with a specific value. The total score ranges from -4 to 12.
  Interpretation:
  ≤3: Very-low-quality diet. 4-7: Need to improve the food pattern to align with the Mediterranean diet.
  ≥8: Optimal adherence to the Mediterranean diet. A lower overall score (≤3) mean a worst outcome (adherence); while a higher overall score (≥8) mean a better outcome (adherence).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: index
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
index | 6.37 (2.67) | 5.77 (2.78) | 5.00 (2.00)

25. Secondary Outcome: Mediterranean Diet Index (KIDMED) Analysis
Description: specific foods frequency consumption based on the KIDMED questionnaire
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 30 | 30
Participants
  1 Fruit - fruit juice daily | 16 | 22 | 20
  Fruits daily >2 | 7 | 13 | 12
  1 Fresh - cooked vegetable daily | 18 | 18 | 22
  Fresh - cooked vegetable daily >1 | 6 | 10 | 5
  Fish regularly > 2 per week | 9 | 15 | 16
  Fast food >1 per week | 12 | 5 | 9
  Legumes >1 per week | 20 | 17 | 21
  Pasta - rice daily | 25 | 23 | 23
  Cereals - grains daily | 28 | 29 | 27
  Nuts > 2 times per week | 9 | 14 | 8
  Olive oil daily | 29 | 28 | 29
  Skipping breakfast | 7 | 6 | 9
  Dairy at breakfast | 24 | 25 | 26
  Commercial pastries - pastries at breakfast | 18 | 13 | 16
  2 Yogurt - cheese servings daily | 19 | 18 | 20
  Sweets and candies daily | 23 | 17 | 22

26. Secondary Outcome: Anti-TPOAb
Description: antithyroid peroxidase antibody (Anti-TPOAb) titers
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the baseline and 6 month time points.
Measure: Median (Inter-Quartile Range); unit: IU/mL
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 0 | 0
IU/mL
  baseline | 979.50 [135.27 to 2383.72] |  |
  6 months | 800.00 [73.47 to 1687.20] |  |

27. Secondary Outcome: Anti-TgAb
Description: thyroglobulin antibody (Anti-TgAb) titers
Time Frame: baseline and 6 months
Population: Data have not been collected for the "Control Group" and "AIT Euthyroid Group" for the baseline and 6 month time points.
Measure: Median (Inter-Quartile Range); unit: IU/mL
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
Number analyzed (Participants) | 30 | 0 | 0
IU/mL
  baseline | 283.90 [69.40 to 500.00] |  |
  6 months | 236.20 [87.95 to 500.00] |  |

ADVERSE EVENTS:
Time Frame: 0
Description: All-Cause Mortality, Serious, and Other (Not including Serious) Adverse Events were not monitored/assessed
Groups:
- AIT Subclinical Hypothyroid Group: Children and Adolescents diagnosed with chronic autoimmune thyroiditis (AIT) and subclinical hypothyroidism (SCH)
- Control Group: Healthy individuals with no chronic autoimmune thyroiditis (AIT) and normal thyroid function
- AIT Euthyroid Group: Children and Adolescents diagnosed with chronic autoimmune thyroiditis (AIT) and euthyroidism.
Arm/Group | AIT Subclinical Hypothyroid Group | Control Group | AIT Euthyroid Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No randomization; relative small sample size; serum FGF-21 levels were not measured in AIT euthyroid patients, as previous animal studies revealed that exogenous FGF-21 administration to hypothyroid animal models led to similar serum and liver lipid metabolites and gene expression changes in both hypothyroid and euthyroid mice. Patients did not have severe long-standing hypothyroidism.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-10-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT02725879/Prot_SAP_ICF_000.pdf